CLINICAL TRIAL: NCT05744128
Title: Positron Emission Tomography Repeatability Evaluation of Tissue Zirconium 89Zr Crefmirlimab Berdoxam
Brief Title: CD8 Minibody Repeatability Study
Acronym: PRETZCEL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: ImaginAb, Inc. (Industry)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IAB-CD8-204
Record Dates: First submitted 2023-01-19; First posted 2023-02-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Melanoma; Renal Cell Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Eligible subjects will receive up to two zirconium Zr 89 crefmirlimab berdoxam PET scans (up to 1.0 mCi ± 20% at 1.5 mg API per scan, for a total of up to 2.0 mCi ± 20% and 3.0 mg API) as an IV infusion or slow bolus injection.
  PET/CT imaging is performed 24hrs ± 3hrs post administration. The two scans are performed a minimum 2 weeks apart.
  Interventions: Biological: Zirconium 89Zr crefmirlimab berdoxam

INTERVENTIONS:
Biological: Zirconium 89Zr crefmirlimab berdoxam — Zirconium-89 labelled minibody for whole body PET imaging to visualize CD8+ cell distribution.
  Other Names: Zr-89 Df-crefmirlimab; Zr-89 Df-IAB22M2C

SUMMARY:
Zr-89 crefmirlimab berdoxam is a Zirconium-89 labelled minibody developed by ImaginAb for full body PET imaging of CD8+ cell distribution (CD8 ImmunoPET). The primary objective of this study is to assess the test-retest repeatability of CD8 immunoPET imaging in oncology patients with stable disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* Patients with at least one imageable primary or metastatic lesion > 1 cm in the lymph nodes or soft tissue excluding bone on the most recent standard of care imaging done within the last 3 months
* Cohort 1: Patients with melanoma on single or multiple agent Immune Checkpoint Blockade (ICB) therapy with stable response status following initiation of therapy. Stable disease would be observed over at least 2 consecutive standard of care CT scans (usually done 8-12 weeks apart) after initiation of therapy.
* Cohort 2: Patients with untreated renal cell carcinoma on active surveillance
* Women of child bearing potential must not be pregnant on study entry
* Participants must agree to follow contraceptive advice while on study and for 30 days after ending participation.

Exclusion Criteria:

* Patients with uncontrolled infection or other concurrent malignancies or conditions that may confound interpretation of the scans in the opinion of the investigator
* Patients with urinary catheters or stoma bags
* Patients who have received a vaccine recently can be included to the study but can only be scanned after a washout period of 2 weeks after the vaccine. If participants have a vaccine after the first PET-CT scan, the second PET-CT scan will be delayed for at least 2 weeks after the vaccine
* Patients on steroids except those on replacement dose of steroids for adrenal or pituitary insufficiency. Patients requiring steroids as therapy for an unresolved immune therapy related adverse event will be excluded
* Participants on immunosuppressive medication e.g. cyclosporine, azathioprine, janus kinase inhibitors
* Participant enrolled into another therapeutic intervention study
* Any other contraindication that makes the patient unsuitable to take part in the study in the opinion of the investigator
* Women who are pregnant or breast feeding
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
SUVs in tumor | 2-4 weeks
  Absolute and relative difference in tumor SUVs
SUVs in reference tissues | 2-4 weeks
  Absolute and relative difference in reference tissue SUVs
ratio of tumor SUVs to reference tissue SUVs | 2-4 weeks
  Absolute and relative difference in SUV ratios

SECONDARY OUTCOMES:
Safety of repeat doses of Zr-89 crefmirlimab berdoxam | Through study completion, an average of 8 weeks
  Adverse events collected during the trial and as self-reported events.

CONTACTS AND LOCATIONS:
Overall Officials: Azeem Saleem, MB BS DMRT PhD FRCR, Principal Investigator — Castle Hill Hospital, Hull
Locations (1):
- Castle Hill Hospital, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No